CLINICAL TRIAL: NCT02373904
Title: A Prospective, Multi-Center Study of the IlluminOss Photodynamic Bone Stabilization System for the Treatment of Impending and Actual Pathological Fractures in the Humerus From Metastatic Bone Disease
Brief Title: A Safety and Efficacy Study of the Treatment of Impending and Actual Pathological Fractures in the Humerus From Metastatic Bone Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IlluminOss Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-03-PATHOLHUM-01; NL49653.072.14 (Other: Institutional Review Board Nijmegen)
Record Dates: First submitted 2015-02-17; First posted 2015-02-27 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Humerus Pathological Fracture

ARMS (1):
- Photodynamic Bone Stabilization System (PBSS) (Experimental): The PBSS is comprised of an inflatable, thin walled polyethylene terephthalate (PET; Dacron™) balloon mounted on an insertion catheter. This balloon catheter system is designed to deliver the monomer cement to the fracture site via the medullary canal of the bone.
  Interventions: Device: Photodynamic Bone Stabilization System

INTERVENTIONS:
Device: Photodynamic Bone Stabilization System — Treatment of impending and actual pathological fractures of the humerus

SUMMARY:
The purpose of this study is to collect safety and performance data of the Photodynamic Bone Stabilization System (PBSS) when used for the treatment of painful impending and actual fractures of the humerus secondary to metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

-General Inclusion Criteria

1. Skeletally mature adult males and females 18 years of age or older.
2. Impending or actual pathological fracture of the humerus, secondary to metastatic bone disease.
3. Females: neither pregnant nor intending to become pregnant during the course of the study, defined as:

   1. Postmenopausal for at least 1 year OR
   2. Documented oophorectomy or hysterectomy
   3. Surgically sterile OR
   4. If of childbearing potential, must be practicing double-barrier method of birth control, be willing to avoid pregnancy for the period of study participation and have a negative pregnancy test at screening
4. Able to understand and provide informed consent.
5. Willing and able to comply with post-operative treatment protocol and follow-up visit schedule.

   -Impending Fracture-Specific Inclusion Criteria
6. Documented presence of solitary metastatic lesion.
7. Mirels Criteria Score ≥ 8.
8. Destruction of cortical bone at impending fracture site > 50%.

   -Actual Fracture-Specific Inclusion Criteria
9. Radiograph-confirmed diagnosis of acute, single isolated fracture of the humerus. AO classification 11A1, 11A2 and 11B1, 11B2 and 12A1,12A2 and 12B1, 12B2 and 13A1,13A2 and 13B1, 13B2.
10. Fracture is closed, Gustilo Type I or IIA.

Exclusion Criteria:

-General Exclusion Criteria

1. Primary tumor (osteogenic origin, etc.) at site.
2. Impending fracture or actual fracture location other than humerus.
3. Current concomitant traumatic fracture of any other location.
4. Active or incompletely treated infections that could involve the device implant site.
5. Distant foci of infection that may spread to the implant site.
6. Allergy to implant materials or dental glue.
7. Vascular insufficiency, muscular atrophy, or neuromuscular disease at implant site.
8. Uncooperative patients, or patients who are incapable of following directions (for example, as a consequence of a neurological or psychiatric disorder).

   -Impending Fracture-Specific Exclusion Criteria
9. Mirels Score < 8.
10. Destruction of cortical bone at impending fracture site < 50%.
11. Prior surgery and/or prior fracture of affected site.
12. Any articular component to impending fracture site.

    -Actual Fracture-Specific Exclusion Criteria
13. Index treatment is greater than 28 days post fracture.
14. Open fractures with severe contamination.
15. Extremely comminuted fractures where insufficient holding power of the balloon on the intramedullary canal is probable.
16. Delivery sheath is unable to cross fracture site after proper fracture reduction and realignment
17. Patients whose intramedullary canal at site of fracture measures smaller than the diameter of the sheath provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | 90 days
  VAS Pain Score change of > -33% compared to baseline
Functional Improvement (Barthel Index of Activities of Daily Living (ADLs) improvement of > +10% from baseline -EORTC QLQ-C30 improvement of > +10% from baseline -EORTC QLQ-BM22 improvement of > +10% from baseline) | 90 days
  * Barthel Index of Activities of Daily Living (ADLs) improvement of > +10% from baseline
  * EORTC QLQ-C30 improvement of > +10% from baseline
  * EORTC QLQ-BM22 improvement of > +10% from baseline
Clinical Safety Success (No Serious Device Related Complications -No additional surgical interventions: revisions, supplements, fixations or removals) | 90 days
  * No Serious Device Related Complications
  * No additional surgical interventions: revisions, supplements, fixations or removals
Radiographic Safety Success (No device fracture, migrations, mal-alignment or loss of reduction or fixation) | 90 days
  No device fracture, migrations, mal-alignment or loss of reduction or fixation

SECONDARY OUTCOMES:
Pain Reduction (VAS Pain Score change of > -33% compared to baseline) | 90, 180 and 360 days
  VAS Pain Score change of > -33% compared to baseline
Functional Improvement (-Barthel Index of Activities of Daily Living (ADLs) improvement of > +10% from baseline, -EORTC QLQ-C30 improvement of > +10% from baseline -EORTC QLQ-BM22 improvement of > +10% from baseline) | 90, 180, 360 days
  * Barthel Index of Activities of Daily Living (ADLs) improvement of > +10% from baseline,
  * EORTC QLQ-C30 improvement of > +10% from baseline
  * EORTC QLQ-BM22 improvement of > +10% from baseline
Clinical Safety Success (No Serious Device Related Complications -No additional surgical interventions: revisions, supplements, fixations or removals) | 90, 180, 360 days
  * No Serious Device Related Complications
  * No additional surgical interventions: revisions, supplements, fixations or removals
Radiographic Safety Success (No device fracture, migrations, mal-alignment or loss of reduction or fixation) | 90, 180, 360 days
  No device fracture, migrations, mal-alignment or loss of reduction or fixation
Duration of index procedure and length of hospital stay | 90, 180, 360 days
Disability status | 90, 180, 360 days
  Determined per Investigator assessment
Evaluation of duration of physical therapy prescription | 90, 180, 360 days
Assessment of prescription and over-the-counter analgesic medication use | 90, 180, 360 days
Survivability from time of index procedure to death | 90, 180, 360 days
Incidence and number of AEs | 90, 180, 360 days
Incidence and number of procedure- and device-related complications | 90, 180, 360 days
Activities of Daily Living score through all follow-up intervals | 90, 180, 360 days
  Barthel Index of Activities of Daily Living (ADLs), EORTC QLQ-C30 and EORTC QLQ-BM22
VAS Pain score from baseline through all follow-up intervals | 90, 180, 360 days
  VAS pain scale

CONTACTS AND LOCATIONS:
Locations (6):
- Medical University of Vienna, Vienna, Austria
- Germany (3):
  - St. Vinzenz-Hospital GmbH, Cologne
  - Johannes Wesling Klinikum Minden, Minden
  - Lahn-Dill Kliniken, Wetzlar
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede
  - Medical Center Leeuwarden, Leeuwarden